CLINICAL TRIAL: NCT04650750
Title: The Treatment Effect of Chinese Medicine Formula on Uremic Pruritus
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMRPG1J0131
Record Dates: First submitted 2020-10-28; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-10

CONDITIONS: Uremic Pruritus
Keywords: Uremic pruritus; Hemodialysis; Chinese medicine; Xiao-Feng-San; Shian Fang Hwa Ming Yiin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xiao-Feng-San; Shian-Fang-Hwa-Ming-Yiin (Experimental): Xiao-Feng-San 2g+ Shian Fang Hwa Ming Yiin 2g; twice a day for two months
  Interventions: Drug: Xiao-Feng-San+Shian-Fang-Hwa-Ming-Yiin
- Placebo (Placebo Comparator): Similar placebo 4g twice a day for two months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xiao-Feng-San+Shian-Fang-Hwa-Ming-Yiin — "Xiao-Feng-San" is a common Chinese herbal preparation, composed of 13 herbs, which is used to treat patients with dermatitis. The component of "Xiao-Feng-San" has immunomodulatory activity. "Shian Fang Hwa Ming Yiin" is another common Chinese herbal preparation, composed of 12 herbs, which is used to treat patients with carbuncles and acne. The component of "Shian Fang Hwa Ming Yiin" has anti-inflammation and anti-microbial effect.
  Arms: Xiao-Feng-San; Shian-Fang-Hwa-Ming-Yiin
Drug: Placebo — Similar placebo 4g twice a day for two months
  Arms: Placebo

SUMMARY:
The prevalence of hemodialysis patients is increasing in recent years. And the uremic pruritus is a common and bothersome symptom among the patients. Current therapies for uremic pruritus, including dialysis modification, topical treatment such as emollients and topical analgesic agent, phototherapy, acupuncture, and gabapentin. However, the efficacy of these treatments remains poorly defined.

In our experiment, the investigators tried to find an effective way to control uremic pruritus through Chinese traditional medicine.

DETAILED DESCRIPTION:
The prevalence of hemodialysis patients is increasing in recent years. And the uremic pruritus is a common and bothersome symptom among the patients. Current therapies for uremic pruritus, including dialysis modification, topical treatment such as emollients and topical analgesic agent, phototherapy, acupuncture, and gabapentin. However, the efficacy of these treatments remains poorly defined.

In our experiment, the investigators tried to find an effective way to control uremic pruritus through Chinese traditional medicine. "Xiao-Feng-San" is a common Chinese herbal preparation, composed of 13 herbs, which is used to treat patients with dermatitis. The component of "Xiao-Feng-San" has immunomodulatory activity. "Shian Fang Hwa Ming Yiin" is another common Chinese herbal preparation, composed of 12 herbs, which is used to treat patients with carbuncles and acne. The component of "Shian Fang Hwa Ming Yiin" has anti-inflammation and anti-microbial effect.

The purpose of this study is to evaluate the treatment effect of Xiao-Feng-San and Shian Fang Hwa Ming Yiin on uremic pruritus among hemodialysis patients in this randomized, double-blind, placebo-controlled study design.

ELIGIBILITY:
Inclusion Criteria:

1. At least 3 episodes of itch during 2 weeks or less, the itch occurring several times a day, lasting for more than 5 min and being bothersome
2. An intermittent itch over a period of 6 months or more, with a clinical appearance, but with a lower frequency than in (1)
3. People with clear consciousness, without cognitive impairment
4. Those who can cooperate to fill in relevant questionnaires
5. Willing to sign consent forms
6. Blood test indicators: (1) Intact parathyroid hormone (iPTH) <600 pg/ml (2) Kt/V >1.2 (3) Serum phosphate <6 mg/dl
7. Refractory uremic pruritus; The patient failed to respond to following treatments (1) avoiding food containing high amounts of phosphate (2) haemodialysis with a dialysate containing 3.0 or 2.5 mEq/l of calcium (3) changing the dialyser or increasing blood flow

Exclusion Criteria:

1. Be younger than 20 years old.
2. People suffering from diagnosed skin diseases (scabies, drug allergy, atopic dermatitis), severe infections, liver failure, blood diseases or biliary diseases.
3. Patients with abnormal liver and kidney function.
4. People suffering from cognitive dysfunction caused by neurological diseases or mental diseases.
5. People with severe visual impairment, hearing impairment, and physical impairment that affect the scale test.
6. Those who are undergoing other trials.
7. Those who are pregnant or breastfeeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale(VAS) | on starting day (day 0)
  Measuring itch intensity
Visual Analogue Scale(VAS) | on day 28
  Measuring itch intensity
Visual Analogue Scale(VAS) | on day 56
  Measuring itch intensity
Visual Analogue Scale(VAS) | on day 84
  Measuring itch intensity
5-D itch scale | on starting day (day 0)
  (1) duration of itchiness, (2) degree of itchiness, (3) direction of itchiness, (4) disability caused by itchiness, and (5) distribution of itchiness
5-D itch scale | on day 28
  (1) duration of itchiness, (2) degree of itchiness, (3) direction of itchiness, (4) disability caused by itchiness, and (5) distribution of itchiness
5-D itch scale | on day 56
  (1) duration of itchiness, (2) degree of itchiness, (3) direction of itchiness, (4) disability caused by itchiness, and (5) distribution of itchiness
5-D itch scale | on day 84
  (1) duration of itchiness, (2) degree of itchiness, (3) direction of itchiness, (4) disability caused by itchiness, and (5) distribution of itchiness

REFERENCES:
- [Background] Mathur VS, Lindberg J, Germain M, Block G, Tumlin J, Smith M, Grewal M, McGuire D; ITCH National Registry Investigators. A longitudinal study of uremic pruritus in hemodialysis patients. Clin J Am Soc Nephrol. 2010 Aug;5(8):1410-9. doi: 10.2215/CJN.00100110. Epub 2010 Jun 17. PMID 20558560
- [Background] Rayner HC, Larkina M, Wang M, Graham-Brown M, van der Veer SN, Ecder T, Hasegawa T, Kleophas W, Bieber BA, Tentori F, Robinson BM, Pisoni RL. International Comparisons of Prevalence, Awareness, and Treatment of Pruritus in People on Hemodialysis. Clin J Am Soc Nephrol. 2017 Dec 7;12(12):2000-2007. doi: 10.2215/CJN.03280317. Epub 2017 Sep 18. PMID 28923831
- [Background] Kuypers DR. Skin problems in chronic kidney disease. Nat Clin Pract Nephrol. 2009 Mar;5(3):157-70. doi: 10.1038/ncpneph1040. Epub 2009 Feb 3. PMID 19190625
- [Background] Szepietowski JC, Morita A, Tsuji T. Ultraviolet B induces mast cell apoptosis: a hypothetical mechanism of ultraviolet B treatment for uraemic pruritus. Med Hypotheses. 2002 Feb;58(2):167-70. doi: 10.1054/mehy.2001.1505. PMID 11812197
- [Background] Kim KH, Lee MS, Choi SM. Acupuncture for treating uremic pruritus in patients with end-stage renal disease: a systematic review. J Pain Symptom Manage. 2010 Jul;40(1):117-25. doi: 10.1016/j.jpainsymman.2009.11.325. PMID 21796811
- [Background] Okada K, Matsumoto K. Effect of skin care with an emollient containing a high water content on mild uremic pruritus. Ther Apher Dial. 2004 Oct;8(5):419-22. doi: 10.1111/j.1526-0968.2004.00175.x. PMID 15663539
- [Background] Young TA, Patel TS, Camacho F, Clark A, Freedman BI, Kaur M, Fountain J, Williams LL, Yosipovitch G, Fleischer AB Jr. A pramoxine-based anti-itch lotion is more effective than a control lotion for the treatment of uremic pruritus in adult hemodialysis patients. J Dermatolog Treat. 2009;20(2):76-81. doi: 10.1080/09546630802441218. PMID 18821119
- [Background] Tarng DC, Cho YL, Liu HN, Huang TP. Hemodialysis-related pruritus: a double-blind, placebo-controlled, crossover study of capsaicin 0.025% cream. Nephron. 1996;72(4):617-22. doi: 10.1159/000188949. PMID 8730431
- [Background] Russo GE, Spaziani M, Guidotti C, Scarpellini MG, Leri O, Bonini S, Crisciotti C, Carmenini G. [Pruritus in chronic uremic patients in periodic hemodialysis. Treatment with terfenadine (an antagonist of histamine H1 receptors)]. Minerva Urol Nefrol. 1986 Oct-Dec;38(4):443-7. No abstract available. Italian. PMID 2884733
- [Background] Rayner H, Baharani J, Smith S, Suresh V, Dasgupta I. Uraemic pruritus: relief of itching by gabapentin and pregabalin. Nephron Clin Pract. 2012;122(3-4):75-9. doi: 10.1159/000349943. Epub 2013 Mar 28. PMID 23548570
- [Background] Simonsen E, Komenda P, Lerner B, Askin N, Bohm C, Shaw J, Tangri N, Rigatto C. Treatment of Uremic Pruritus: A Systematic Review. Am J Kidney Dis. 2017 Nov;70(5):638-655. doi: 10.1053/j.ajkd.2017.05.018. Epub 2017 Jul 15. PMID 28720208
- [Background] Cheng HM, Chiang LC, Jan YM, Chen GW, Li TC. The efficacy and safety of a Chinese herbal product (Xiao-Feng-San) for the treatment of refractory atopic dermatitis: a randomized, double-blind, placebo-controlled trial. Int Arch Allergy Immunol. 2011;155(2):141-8. doi: 10.1159/000318861. Epub 2010 Dec 22. PMID 21196758
- [Background] Chen HY, Lin YH, Chen YC. Identifying Chinese herbal medicine network for treating acne: Implications from a nationwide database. J Ethnopharmacol. 2016 Feb 17;179:1-8. doi: 10.1016/j.jep.2015.12.032. Epub 2015 Dec 22. PMID 26721214